CLINICAL TRIAL: NCT00310726
Title: Short Duration Exclusive Breastfeeding With Abrupt Weaning to Reduce the Risk of Mother-to-Child HIV Transmission
Brief Title: Zambia Exclusive Breastfeeding Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Donald M. Thea, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD039611 (NIH); R01HD039611 (NIH)
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: HIV Infection
Keywords: Mother to Child Transmission of HIV; Postnatal HIV transmission; HIV; Breastfeeding; Perinatal HIV Transmission; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abrupt Weaning (Experimental): Women were counseled to abruptly wean their child at 4 months of age.
  Interventions: Other: abrupt weaning at 4 months
- Exclusive breastfeeding per WHO guidelines (Active Comparator): Women were counseled to adhere to the WHO recommendations for duration of exclusive breastfeeding.
  Interventions: Other: Continued exclusive breastfeeding

INTERVENTIONS:
Other: abrupt weaning at 4 months — abrupt weaning at 4 months
  Arms: Abrupt Weaning
Other: Continued exclusive breastfeeding — Continued exclusive breastfeeding
  Arms: Exclusive breastfeeding per WHO guidelines

SUMMARY:
The study is designed as a randomized, controlled trial with specific observational objectives. All HIV-seropositive pregnant subjects electing to breastfeed their child will be counselled to exclusively breastfeed through 4 months of age. All live-born children will be randomized (1:1) at birth to one of two counseling programs: A) to encourage abrupt weaning at 4 months of age, or B) to encourage exclusive breastfeeding through 6 months of age with the introduction of typical weaning foods ad lib.

DETAILED DESCRIPTION:
It is well established that infants breast fed by their HIV-infected mothers are at risk of acquiring HIV infection through breast milk. However, in low resource settings, where the HIV epidemic now predominates, breast feeding cannot simply be replaced by breast milk substitutes since alternatives to breast milk are unavailable, unaffordable and unsafe. With this application we aim to test the safety and efficacy of short duration exclusive breast feeding to minimize risks of HIV transmission without increasing risks of non-HIV infant mortality. We propose a 5-year study of HIV-positive mothers and their children to be conducted in two urban primary health care clinics in Lusaka, Zambia. All HIV-positive women and their infants will be offered the two-dose nevirapine intervention and will be counseled about the risks and benefits of infant feeding options. Women who indicate their decision to breast feed will be eligible for enrollment into the study. A culturally appropriate, affordable and sustainable breast feeding education and support program to encourage exclusive breast feeding will be developed, and all women who elect to breast feed will be encouraged to exclusively breast feed to 4 months. Half of the women will be randomized to a counseling program which will encourage abrupt weaning to full replacement feeding at 4 months, and half will be randomized to a program to encourage continued breast feeding after 4 months with the usual introduction of weaning foods. Children will be followed for two years with regular medical histories, physical exams and clinical sampling. The primary objective of the study, based on the random assignment, is to compare HIV transmission rates and under-2 year mortality rates in children who abruptly wean at four months of age versus children who are weaned according to local practice. The second primary objective, based on observational comparisons, is to compare HIV transmission among infants whose mothers adhere to recommendations to exclusively breast feed with those who do not. Secondary objectives are to describe acute and chronic effects of abrupt weaning on child morbidity. The study proposes to test an inexpensive and potentially sustainable public health intervention to reduce HIV transmission through breast feeding while preserving benefits of breast feeding for other aspects of child health in a very low resource setting.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive pregnant women identified through VCT
* After counseling about the risks and benefits of feeding alternatives report that it is their intended decision to breastfeed
* Live within the catchment area of George or Chawama clinic
* Are between 30 - 34 wks gestation. (To insure that opportunity exists to receive a minimum of 2 lactation counseling sessions prior to delivery)
* Do not have any significant presenting illness that requires hospitalization
* Agree to adhere to the requirements of study participation (including exclusive breastfeeding and randomization into one of two infant feeding groups at four months).
* Willing to inform a household member (preferably husband/father) of HIV-status.

Exclusion Criteria:

* Lives outside of catchment area;
* Have known major illnesses likely to influence pregnancy outcome including diabetes, severe renal or heart disease, or active tuberculosis, prior to randomization;
* Does not intend to breastfeed;
* Prior enrollment in this study or concurrent enrollment in another study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1435 (Actual)
Dates: Start 2001-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HIV infection detected by 4 months among children with no evidence of HIV infection at birth. | 24 months of age
Magnitude of the reduction in mother-to-child HIV transmission and the magnitude of the increase in non-HIV-related under-2-year mortality, attributable to cessation of breastfeeding at 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kuhn, PhD, Principal Investigator — Gertrude H. Sergievsky Center, and Department of Epidemiology, Mailman School of Public Health, Columbia University; Donald M Thea, MD, MSc, Principal Investigator — Department of International Health, Boston University School of Public Health
Locations (1):
- George and Chawama District Health Clinics, Lusaka, Zambia

REFERENCES:
- [Background] Thea DM, Vwalika C, Kasonde P, Kankasa C, Sinkala M, Semrau K, Shutes E, Ayash C, Tsai WY, Aldrovandi G, Kuhn L. Issues in the design of a clinical trial with a behavioral intervention--the Zambia exclusive breast-feeding study. Control Clin Trials. 2004 Aug;25(4):353-65. doi: 10.1016/j.cct.2004.06.005. PMID 15296810
- [Background] Kuhn L, Aldrovandi GM, Sinkala M, Kankasa C, Mwiya M, Thea DM. Potential impact of new WHO criteria for antiretroviral treatment for prevention of mother-to- child HIV transmission. AIDS. 2010 Jun 1;24(9):1374-7. PMID 20568677
- [Result] Albrecht S, Semrau K, Kasonde P, Sinkala M, Kankasa C, Vwalika C, Aldrovandi GM, Thea DM, Kuhn L. Predictors of nonadherence to single-dose nevirapine therapy for the prevention of mother-to-child HIV transmission. J Acquir Immune Defic Syndr. 2006 Jan 1;41(1):114-8. doi: 10.1097/01.qai.0000179425.27036.d7. PMID 16340483
- [Result] Kuhn L, Kasonde P, Sinkala M, Kankasa C, Semrau K, Scott N, Tsai WY, Vermund SH, Aldrovandi GM, Thea DM. Does severity of HIV disease in HIV-infected mothers affect mortality and morbidity among their uninfected infants? Clin Infect Dis. 2005 Dec 1;41(11):1654-61. doi: 10.1086/498029. Epub 2005 Oct 27. PMID 16267740
- [Result] Kuhn L, Kasonde P, Sinkala M, Kankasa C, Semrau K, Vwalika C, Tsai WY, Aldrovandi GM, Thea DM. Prolonged breast-feeding and mortality up to two years post-partum among HIV-positive women in Zambia. AIDS. 2005 Oct 14;19(15):1677-81. doi: 10.1097/01.aids.0000186817.38112.da. PMID 16184038
- [Result] Kuhn L, Trabattoni D, Kankasa C, Semrau K, Kasonde P, Lissoni F, Sinkala M, Ghosh M, Vwalika C, Aldrovandi GM, Thea DM, Clerici M. Alpha-defensins in the prevention of HIV transmission among breastfed infants. J Acquir Immune Defic Syndr. 2005 Jun 1;39(2):138-42. PMID 15905728
- [Result] Semrau K, Kuhn L, Vwalika C, Kasonde P, Sinkala M, Kankasa C, Shutes E, Aldrovandi G, Thea DM. Women in couples antenatal HIV counseling and testing are not more likely to report adverse social events. AIDS. 2005 Mar 24;19(6):603-9. doi: 10.1097/01.aids.0000163937.07026.a0. PMID 15802979
- [Result] Ghosh MK, Kuhn L, West J, Semrau K, Decker D, Thea DM, Aldrovandi GM. Quantitation of human immunodeficiency virus type 1 in breast milk. J Clin Microbiol. 2003 Jun;41(6):2465-70. doi: 10.1128/JCM.41.6.2465-2470.2003. PMID 12791866
- [Result] Sabbaj S, Edwards BH, Ghosh MK, Semrau K, Cheelo S, Thea DM, Kuhn L, Ritter GD, Mulligan MJ, Goepfert PA, Aldrovandi GM. Human immunodeficiency virus-specific CD8(+) T cells in human breast milk. J Virol. 2002 Aug;76(15):7365-73. doi: 10.1128/jvi.76.15.7365-7373.2002. PMID 12097549
- [Result] Fawzy A, Arpadi S, Kankasa C, Sinkala M, Mwiya M, Thea DM, Aldrovandi GM, Kuhn L. Early weaning increases diarrhea morbidity and mortality among uninfected children born to HIV-infected mothers in Zambia. J Infect Dis. 2011 May 1;203(9):1222-30. doi: 10.1093/infdis/jir019. PMID 21459815
- [Result] Gray RR, Salemi M, Lowe A, Nakamura KJ, Decker WD, Sinkala M, Kankasa C, Mulligan CJ, Thea DM, Kuhn L, Aldrovandi G, Goodenow MM. Multiple independent lineages of HIV-1 persist in breast milk and plasma. AIDS. 2011 Jan 14;25(2):143-52. doi: 10.1097/QAD.0b013e328340fdaf. PMID 21173592
- [Result] Murnane PM, Arpadi SM, Sinkala M, Kankasa C, Mwiya M, Kasonde P, Thea DM, Aldrovandi GM, Kuhn L. Lactation-associated postpartum weight changes among HIV-infected women in Zambia. Int J Epidemiol. 2010 Oct;39(5):1299-310. doi: 10.1093/ije/dyq065. Epub 2010 May 19. PMID 20484334
- [Result] Heath L, Conway S, Jones L, Semrau K, Nakamura K, Walter J, Decker WD, Hong J, Chen T, Heil M, Sinkala M, Kankasa C, Thea DM, Kuhn L, Mullins JI, Aldrovandi GM. Restriction of HIV-1 genotypes in breast milk does not account for the population transmission genetic bottleneck that occurs following transmission. PLoS One. 2010 Apr 20;5(4):e10213. doi: 10.1371/journal.pone.0010213. PMID 20422033
- [Result] Kuhn L, Sinkala M, Semrau K, Kankasa C, Kasonde P, Mwiya M, Hu CC, Tsai WY, Thea DM, Aldrovandi GM. Elevations in mortality associated with weaning persist into the second year of life among uninfected children born to HIV-infected mothers. Clin Infect Dis. 2010 Feb 1;50(3):437-44. doi: 10.1086/649886. PMID 20047479
- [Result] Walter J, Ghosh MK, Kuhn L, Semrau K, Sinkala M, Kankasa C, Thea DM, Aldrovandi GM. High concentrations of interleukin 15 in breast milk are associated with protection against postnatal HIV transmission. J Infect Dis. 2009 Nov 15;200(10):1498-502. doi: 10.1086/644603. PMID 19835475
- [Result] Walter J, Kuhn L, Semrau K, Decker DW, Sinkala M, Kankasa C, Thea DM, Bulterys M, Ou CY, Aldrovandi GM. Detection of low levels of human immunodeficiency virus (HIV) may be critical for early diagnosis of pediatric HIV infection by use of dried blood spots. J Clin Microbiol. 2009 Sep;47(9):2989-91. doi: 10.1128/JCM.02453-08. Epub 2009 Jul 22. PMID 19625479
- [Result] Kuhn L, Aldrovandi GM, Sinkala M, Kankasa C, Semrau K, Kasonde P, Mwiya M, Tsai WY, Thea DM; Zambia Exclusive Breastfeeding Study (ZEBS). Differential effects of early weaning for HIV-free survival of children born to HIV-infected mothers by severity of maternal disease. PLoS One. 2009 Jun 26;4(6):e6059. doi: 10.1371/journal.pone.0006059. PMID 19557167
- [Result] Arpadi S, Fawzy A, Aldrovandi GM, Kankasa C, Sinkala M, Mwiya M, Thea DM, Kuhn L. Growth faltering due to breastfeeding cessation in uninfected children born to HIV-infected mothers in Zambia. Am J Clin Nutr. 2009 Aug;90(2):344-53. doi: 10.3945/ajcn.2009.27745. Epub 2009 Jun 24. PMID 19553300
- [Result] Kuhn L, Semrau K, Ramachandran S, Sinkala M, Scott N, Kasonde P, Mwiya M, Kankasa C, Decker D, Thea DM, Aldrovandi GM. Mortality and virologic outcomes after access to antiretroviral therapy among a cohort of HIV-infected women who received single-dose nevirapine in Lusaka, Zambia. J Acquir Immune Defic Syndr. 2009 Sep 1;52(1):132-6. doi: 10.1097/QAI.0b013e3181ab6d5e. PMID 19506483
- [Result] Walter J, Kuhn L, Kankasa C, Semrau K, Sinkala M, Thea DM, Aldrovandi GM. Reuse of single-dose nevirapine in subsequent pregnancies for the prevention of mother-to-child HIV transmission in Lusaka, Zambia: a cohort study. BMC Infect Dis. 2008 Dec 30;8:172. doi: 10.1186/1471-2334-8-172. PMID 19116004
- [Result] Fox MP, Brooks DR, Kuhn L, Aldrovandi G, Sinkala M, Kankasa C, Horsburgh R, Thea DM. Role of breastfeeding cessation in mediating the relationship between maternal HIV disease stage and increased child mortality among HIV-exposed uninfected children. Int J Epidemiol. 2009 Apr;38(2):569-76. doi: 10.1093/ije/dyn249. Epub 2008 Nov 30. PMID 19047077
- [Result] Kuhn L, Aldrovandi GM, Sinkala M, Kankasa C, Semrau K, Mwiya M, Kasonde P, Scott N, Vwalika C, Walter J, Bulterys M, Tsai WY, Thea DM; Zambia Exclusive Breastfeeding Study. Effects of early, abrupt weaning on HIV-free survival of children in Zambia. N Engl J Med. 2008 Jul 10;359(2):130-41. doi: 10.1056/NEJMoa073788. Epub 2008 Jun 4. PMID 18525036
- [Result] Semrau K, Ghosh M, Kankasa C, Sinkala M, Kasonde P, Mwiya M, Thea DM, Kuhn L, Aldrovandi GM. Temporal and lateral dynamics of HIV shedding and elevated sodium in breast milk among HIV-positive mothers during the first 4 months of breast-feeding. J Acquir Immune Defic Syndr. 2008 Mar 1;47(3):320-8. doi: 10.1097/qai.0b013e31815e7436. PMID 18398972
- [Result] Fox MP, Brooks D, Kuhn L, Aldrovandi G, Sinkala M, Kankasa C, Mwiya M, Horsburgh R, Thea DM. Reduced mortality associated with breast-feeding-acquired HIV infection and breast-feeding among HIV-infected children in Zambia. J Acquir Immune Defic Syndr. 2008 May 1;48(1):90-6. doi: 10.1097/QAI.0b013e31816e39a3. PMID 18344878
- [Result] Kuhn L, Sinkala M, Kankasa C, Semrau K, Kasonde P, Scott N, Mwiya M, Vwalika C, Walter J, Tsai WY, Aldrovandi GM, Thea DM. High uptake of exclusive breastfeeding and reduced early post-natal HIV transmission. PLoS One. 2007 Dec 26;2(12):e1363. doi: 10.1371/journal.pone.0001363. PMID 18159246
- [Result] Castelletti E, Lo Caputo S, Kuhn L, Borelli M, Gajardo J, Sinkala M, Trabattoni D, Kankasa C, Lauri E, Clivio A, Piacentini L, Bray DH, Aldrovandi GM, Thea DM, Veas F, Nebuloni M, Mazzotta F, Clerici M. The mucosae-associated epithelial chemokine (MEC/CCL28) modulates immunity in HIV infection. PLoS One. 2007 Oct 3;2(10):e969. doi: 10.1371/journal.pone.0000969. PMID 17912348
- [Derived] Celerino da Silva R, Segat L, Kuhn L, Chies JAB, Crovella S. Association of SNPs in HLA-C and ZNRD1 Genes With HIV-1 Mother-to-Child Transmission in Zambia Population. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):509-515. doi: 10.1097/QAI.0000000000002584. PMID 33252547
- [Derived] Bode L, Kuhn L, Kim HY, Hsiao L, Nissan C, Sinkala M, Kankasa C, Mwiya M, Thea DM, Aldrovandi GM. Human milk oligosaccharide concentration and risk of postnatal transmission of HIV through breastfeeding. Am J Clin Nutr. 2012 Oct;96(4):831-9. doi: 10.3945/ajcn.112.039503. Epub 2012 Aug 15. PMID 22894939